CLINICAL TRIAL: NCT06718673
Title: The Effect of Virtual Delivery Room Visits on Primiparous Women's Beliefs About Normal Birth and Their Birth Adaptation
Brief Title: The Effect of Virtual Delivery Room Visit on Birth Belief and Adaptation
Acronym: EVDRVBBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Merve AKINCI, Assistant Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-25403353-050.99-294113
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy; Birth; Delivery Room; Midwifery; Virtual Reality; Adaptation
Keywords: Pregnancy; Normal Birth; Birth Adaptation; Normal Birth Tendency.; Virtual Reality; Midwifery; Delivery room

STUDY DESIGN:
Masking Description: Due to the nature of the intervention, it was not possible to blind participants or care providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- virtual delivery room visit (Experimental): Participants were informed about the study, the Participant Information Form was provided during the initial interview, and the Belief Scale for Normal Delivery pre-test was administered. Following, participants in the intervention group were provided with a link to a virtual delivery room introduction video (https://www.youtube.com/watch?v=EyCt-jTDCVs), created using the actual delivery room environment, and were encouraged to watch it., a second interview was conducted four days after the initial interview, during which post-test data were collected using the Belief Scale for Normal Delivery form. After all participants completed their birth processes, a third interview was conducted, and the data collection process was finalized using the Birth Adaptation Self-Assessment Scale and Birth Adaptation Midwife Assessment Scale forms.
  Interventions: Other: virtual delivery room visit
- Standard of care (Other): Participants were informed about the study, the Participant Information Form was provided during the initial interview, and the Belief Scale for Normal Delivery pre-test was administered. However, no intervention related to the virtual delivery room visit was conducted with the control group. This group was only subjected to a monitoring process after the pre-test. Four days after the initial interview, a second interview was conducted with participants in the control group, during which post-test data were collected using the BSND form. After the birth processes of the participants in the control group were completed, a third interview was conducted, and the data collection process was completed using the Birth Adaptation Self-Assessment Scale and Birth Adaptation Midwife Assessment Scale forms.
  Interventions: Other: standart of care

INTERVENTIONS:
Other: virtual delivery room visit — The real-time labour room demonstration video aims to increase participants' awareness of the labour process, reduce unfamiliarity, and facilitate participation for pregnant women with access restrictions. Produced with a 360-degree camera, it shows detailed sections of the labour room, starting from the entrance. Key areas like birthing beds, toilets, bathrooms, and labour materials (mats, pilates balls, TVs) are highlighted. The video also covers baby cots and rest areas for attendants. Narrated by an experienced midwife, the video ensures patient privacy, no interventions, and excludes images or sounds of other pregnant women. Converted to 360-degree format, the video is available on YouTube for repeated viewing. (https://www.youtube.com/watch?v=EyCt-jTDCVs)
  Arms: virtual delivery room visit
Other: standart of care — Pregnant women in the control group did not receive any intervention other than routine care and counselling.
  Arms: Standard of care

SUMMARY:
Aims: The aim is to examine the effect of virtual delivery room visits on primiparous women's beliefs about normal birth and their birth adaptation.

Method: A prospective, randomized controlled study was conducted between July and November 2023 at a training hospital in the Western Black Sea Region of Türkiye. Eighty pregnant women were randomly assigned to the intervention (n=40) and control (n=40) groups. Pre-test data were collected using the Participant Information Form and the Belief Scale for Normal Delivery(BSND), and post-test data were collected with BSND after the virtual delivery room visit. The Birth Adaptation Self-Assessment Scale(BASAS) and Birth Adaptation Midwife Assessment Scale(BAMAS) were administered to the intervention group.

DETAILED DESCRIPTION:
One of the important factors of fear of birth is the uncertainty of pregnant women about the birth environment. Especially primiparous women experience intense fear and anxiety due to insufficient information about the birth process and environment. This situation may negatively affect their birth experience by increasing their level of fear before birth. Birth adaptation refers to a woman's ability to physically and emotionally interact with her environment in a healthy way during the birth process. This adaptation is made possible by women's healthy behaviours and effective cooperation with the healthcare team. This interaction, which is necessary for a positive birth experience, makes women feel safe and contributes to making the birth process more manageable. In this context, in order to prevent uncertainties about the birth process from negatively affecting birth adaptation, it is important for women to recognise the delivery room, to be adequately informed about the birth process and to provide a reassuring environment. These factors enable women to prepare for the birth process more effectively, increase their confidence in the healthcare team and themselves, and make both the physical and emotional dimensions of birth more manageable.

The best way to prepare effectively for the birth process is to participate in antenatal education programmes. These programmes reduce uncertainty by encouraging pregnant women to learn about the birth process and provide an opportunity to familiarise themselves with the delivery room. Women's knowledge of the birth process facilitates healthy behaviour and effective collaboration with health care staff. This process enables women to participate more effectively in the birth process and contributes to their confidence in themselves and the health care team. In addition, antenatal education helps to prevent unnecessary caesarean sections by strengthening beliefs in normal birth.

Improving the quality and accessibility of antenatal education will make a significant contribution to reducing the high cesarean section rates worldwide. In many countries such as Turkey, caesarean section rates are far above the ideal levels (10-15%) set by the World Health Organisation. These high rates carry serious risks for maternal health and it is an urgent necessity to solve this problem. In this context, qualitative and quantitative improvement of antenatal education will be an important step in reducing caesarean section rates.

Time constraints, transport difficulties, inadequacy of trainings and financial barriers are among the main factors preventing regular participation of pregnant women in antenatal education. The COVID-19 pandemic has increased difficulties in accessing healthcare services, leading to the suspension of face-to-face trainings, which has negatively affected pregnant women's preparation for the birth process. Digital trainings help to overcome these barriers, enabling pregnant women to prepare for labour more effectively. In addition, widespread internet access and the demand for reliable information provide a favourable environment for the development of low-cost and widely accessible applications.

The aim of this study was to examine the effect of virtual delivery room visit on primiparous pregnant women's beliefs about normal birth and birth adjustment. The virtual delivery room visit aims to increase birth adjustment and develop positive beliefs towards normal birth by providing pregnant women with the opportunity to get to know the delivery room.

H0 : Virtual delivery room visits have no effect on primiparous women's beliefs about normal birth and their birth adaptation H1a: Virtual delivery room visits increase primiparous women's levels of belief in normal birth.

H1b: Primiparous women who perform a virtual delivery room visit have higher levels of birth adaptation from their own perspective compared to those who do not perform the visit.

H1c: Primiparous women who perform a virtual delivery room visit have higher levels of birth adaptation from their midwives' perspective compared to those who do not perform the visit.

H1d: There is a relationship between primiparous women's beliefs about normal birth and their birth adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Being a primiparous pregnant woman.
* Being between 24 and 40 weeks of gestation.
* Having no pregnancy-related risk factors.
* Not having visited the delivery room of the hospital where the study was conducted prior to the study.
* Planning to give birth at the same hospital.
* Spending at least three hours in labor during childbirth.
* Having access to an internet-connected device.

Exclusion Criteria:

* Refusal to participate in the research.
* Multiparous pregnancy.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Belief Scale for Normal Delivery (BSND) | 3 months
  assesses pregnant women's beliefs about normal birth. It includes 24 items rated on a five-point Likert scale (1-5), with reverse scoring for the perceived barriers subscale (items 12-17). Scores range from 24 to 120, categorized as low (24-56), medium (57-88), or high (89-120).
Birth Adaptation Self-Assessment Scale (BASAS) | 3 months
  Birth Adaptation Self-Assessment Scale, self-assesses a pregnant woman's birth adaptation from her own perspective. The scale contains two subdimensions and a total of 22 items. The two subdimensions are "Midwife-Pregnant Woman Relationship Adaptation" and "Birth Environment Adaptation." Scoring uses a five-point Likert scale, with 1 representing "Strongly Disagree" and 5 representing "Strongly Agree." Item 11 in the "Midwife-Pregnant Woman Relationship Adaptation" subdimension is reverse-scored; there are no reverse-scored items in the "Birth Environment Adaptation" subdimension.
Birth Adaptation Midwife Assessment Scale | 3 months
  Birth Adaptation Midwife Assessment Scale, evaluates whether pregnant women are adapted during their birth processes from the perspective of the midwife who attended the birth. The scale consists of a single subdimension with 17 items. Scoring uses a five-point Likert scale, with 1 representing "Strongly Disagree" and 5 representing "Strongly Agree." Item 8 is reverse-scored.
Participant Information Form | 3 months
  The form collected socio-demographic information such as age, education level, income status, and obstetric characteristics, including the number of pregnancies, number of live births, the desire for the current pregnancy, and information related to pregnancy and birth. The questionnaire comprised a total of 21 questions

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Karabük, Centre, Turkey (Türkiye)